CLINICAL TRIAL: NCT03263169
Title: A Pragmatic Trial to Evaluate the Impact of Community-based Personalized Care on Quality of Life in Older and Disabled Adults
Brief Title: Community-based Personalized Care and QOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Windsor-Essex Compassionate Care Community (Other)
Collaborators: University of Windsor (Other); McMaster University (Other); University of Western Ontario, Canada (Other); Green Shield Canada Inc. (Industry); Erie St. Clair Local Health Integration Network (LHIN) (Other)
Responsible Party: Sponsor
Other Study IDs: HealthTap-WEPilot
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Aging; Disability or Chronic Disease Leading to Disablement
Keywords: e-health, community networks, pragmatic RCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WE Health Tapestry: Completion of baseline measures then enrolled in a community-based personalized care intervention that consists of four core elements: volunteer support, interprofessional care, technology, social network linkage
  Interventions: Behavioral: Community-based personalized care
- Usual Care: Completion of baseline measures with six-month delayed community-based personalized care intervention: volunteer support, interprofessional care, technology, social network linkage
  Interventions: Behavioral: Community-based personalized care

INTERVENTIONS:
Behavioral: Community-based personalized care — volunteer support, health technology, interprofessional care, social network linkage

SUMMARY:
A pragmatic randomized trial to evaluate the impact of an integrated patient experience and outcome measurement system supported by citizens, caregivers and community through eHealth technology.

The primary research question is: What is the effectiveness of the WECCC approach on quality of life in people aged 65 and older or who self-identify as disabled compared to people not receiving the Health TAPESTRY program?

DETAILED DESCRIPTION:
Secondary research questions include:

1. what is the feasibility of obtaining study measures through routinely collected program participant data and what design adjustments are needed to balance pragmatism and high quality data collection?
2. What are the analytic approaches to be developed to aggregate data from individual participants into meaningful units (e.g. care-team level, organizational level, social network, and geographic area) to inform ongoing adaptation of the components of the intervention?
3. what are the perceptions of knowledge users on the usefulness of comparative effectiveness pragmatic trial evidence?

The project involves using administrative data from the ICES to create outcome measures and feedback systems for communities, and the INSPIRE PHC Unit for expertise in health system integration, care in the community, and knowledge translation.

Inclusion criteria: Seniors (65+) and people who self-identify as having a functional disability. Pilot study sites: 7 municipalities and the city of Windsor in Windsor-Essex County in Ontario. The combined total eligible population in all 8 sites is about 60,000 people, from which a minimum sample of 3000 registered patients and 1000 registered caregivers will be drawn

In Year 1, planned enrolment includes a minimum of 1100 intervention clients from all recruitment methods in the care model intervention, with similar numbers of control and intention to treat clients.

The primary outcomes are quality of life (QOL); perceived health; experience of care, and perceived social connection.

The primary outcomes for caregivers will be quality of life; perceived burden; caregiver perceptions of care; and perceived social connection.

Secondary outcomes for both will include goal attainment, distress management, symptom management, places of care, and health care utilization and costs. In terms of health equity, the investigators will measure the difference between the average/median population quality of life and cost outcomes compared to patients at the bottom income quartiles stratified by risk level. At a systems level, algorithms will be developed and applied to the data collected from participants to provide aggregate organization and system-level reports, co-designed with end users to support them as learning organizations.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

1. are 65 years of age and over
2. have a long-term disability or one or more chronic diseases
3. able to communicate in English OR can provide a formal or informal translator willing to facilitate the participant's involvement

Exclusion Criteria:

Individuals not meeting above criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Seniors who identify with having a functional disability or serious chronic disease; and informal caregivers. Many patients within this broad target population will be at risk of worsening quality of life or escalating health care utilization now or in the future due to aging, disease progression, or unmet health, social or economic needs.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Baseline and then monthly for 24 months
  McGill QoL - patient and family
Perceived health | Baseline and then monthly for 24 months
  EQ-5D-5L - patient

SECONDARY OUTCOMES:
Caregiver Burden 1 | Baseline and then monthly for 24 months
  InterRAI-home care
Caregiver Burden 2 | Baseline and then monthly for 24 months
  Zarit burden interview
Patient experience | Baseline and then monthly for 24 months
  CANHelp Patient
Family experience | Baseline and then monthly for 24 months
  CANHelp Family
Symptom management 1 | Baseline and then monthly for 24 months
  Edmonton Symptom Assessment Scale
Symptom management 2 | Baseline and then monthly for 24 months
  Palliative Performance Scale
Symptom management 3 | Baseline and then monthly for 24 months
  InterRAI-home care
Health services utilization 1 | Baseline and then monthly for 24 months
  hospitalization
Health services utilization 2 | Baseline and then monthly for 24 months
  Emergency care

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PhD, Principal Investigator — McMaster University; Lisa Dolovich, PhD, Principal Investigator — McMaster University; Kathryn Pfaff, PhD, Principal Investigator — University of Windsor
Locations (1):
- Windsor-Essex Compassionate Care Community Program Management Office, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided